CLINICAL TRIAL: NCT06039579
Title: A Randomized, Double-Blind (Sponsor Unblinded), Placebo-Controlled, Phase 2a Trial to Investigate the Antiviral Effect, Safety, Tolerability and Pharmacokinetics of Orally Administered Investigational Capsid Inhibitor Monotherapy in HIV-1 Infected Treatment-Naïve Adults
Brief Title: Proof of Concept Treatment Study of Orally Administered VH4004280 or VH4011499 in HIV-1 Infected Adults
Acronym: CINNAMON
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 218307; 2023-505350-18-00 (Other: EU CT number)
Record Dates: First submitted 2023-08-23; First posted 2023-09-15 (Actual); Results first posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: HIV Infections
Keywords: HIV-1; VH4004280; VH4011499; Treatment Naïve; Phase 2a; Monotherapy
MeSH Terms: conditions — HIV Infections | interventions — Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Part 1a: VH4004280 Dose Level 1 (Experimental): Participants received a single dose of VH4004280 Dose Level 1 (low concentration) on Day 1 (evaluated for a 10-day period). On Day 11, participants switched to an open-label antiretroviral therapy (ART) up to day 39.
  Interventions: Drug: VH4004280; Drug: Antiretroviral therapy
- Part 1a: VH4004280 Dose Level 2 (Experimental): Participants received a single dose of VH4004280 Dose Level 2 (medium concentration) on Day 1 (evaluated for a 10-day period). On Day 11, participants switched to an open-label ART up to day 39.
  Interventions: Drug: VH4004280; Drug: Antiretroviral therapy
- Part 2a: VH4004280 pre-specified dose (Experimental): Participants received a single pre-specified dose of VH4004280 (high concentration) on Day 1 (evaluated for a 10-day period). On Day 11, participants switched to an open-label ART up to day 39.
  Interventions: Drug: VH4004280; Drug: Antiretroviral therapy
- Matching placebo for VH4004280 (Placebo Comparator): Participants received a matching placebo for VH4004280 on Day 1 (evaluated for a 10-day period). On Day 11, participants switched to an open-label ART up to day 39.
  Interventions: Drug: VH4004280 Matching Placebo; Drug: Antiretroviral therapy
- Part 1b: VH4011499 Dose Level 1 (Experimental): Participants received a single dose of VH4011499 Dose Level 1 (low concentration) on Day 1 and Day 6 (evaluated for a 10-day period). On Day 11, participants had the option to switch to an open-label ART up to day 39.
  Interventions: Drug: VH4011499; Drug: Antiretroviral therapy
- Part 1b: VH4011499 Dose Level 2 (Experimental): Participants received a single dose of VH4011499 Dose Level 2 (medium concentration) on Day 1 and Day 6 (evaluated for a 10-day period). On Day 11, participants switched to an open-label ART up to day 39.
  Interventions: Drug: VH4011499; Drug: VH4011499 Matching Placebo; Drug: Antiretroviral therapy
- Part 2b: VH4011499 pre-specified dose (Experimental): Participants received a single pre-specified dose of VH4011499 (high concentration) on Day 1 and Day 6 (evaluated for a 10-day period). On Day 11, participants switched to an open-label ART up to day 39.
  Interventions: Drug: VH4011499; Drug: Antiretroviral therapy
- Matching placebo for VH4011499 (Placebo Comparator): Participants received a matching placebo for VH4011499 on Day 1 and Day 6 (evaluated for a 10-day period). On Day 11, participants switched to an open-label ART up to day 39.
  Interventions: Drug: Antiretroviral therapy

INTERVENTIONS:
Drug: VH4004280 — VH4004280 was administered as tablets orally at Day 1.
  Arms: Part 1a: VH4004280 Dose Level 1; Part 1a: VH4004280 Dose Level 2; Part 2a: VH4004280 pre-specified dose
Drug: VH4011499 — VH4011499 was administered as tablets orally at Day 1 and Day 6.
  Arms: Part 1b: VH4011499 Dose Level 1; Part 1b: VH4011499 Dose Level 2; Part 2b: VH4011499 pre-specified dose
Drug: VH4004280 Matching Placebo — VH4004280 Matching Placebo was administered as tablets orally at Day 1.
  Arms: Matching placebo for VH4004280
Drug: VH4011499 Matching Placebo — VH4011499 Matching Placebo was administered as tablets orally at Day 1 and Day 6.
  Arms: Part 1b: VH4011499 Dose Level 2
Drug: Antiretroviral therapy — Antiretroviral therapy was administered as available and as per investigator's recommendation.

SUMMARY:
The primary purpose of the study is to evaluate the antiviral activity of orally administered VH4004280 and VH4011499 monotherapy over 10 days in human immunodeficiency virus (HIV-1) infected Treatment-Naïve (TN) participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy (other than HIV-1 infection).
* Screening cluster of differentiation-4 (CD4+) T-cell count greater than or equal to (≥)200 cells/microliter (µL).
* Documented HIV-1 infection and Screening plasma HIV-1 RNA ≥3000 copies/milliliter (mL).
* Treatment-naïve: Defined as no antiretroviral therapy received after the diagnosis of HIV-1 infection. Prior use of oral pre-exposure prophylaxis (PreP) is permitted. Prior use of parenteral PreP is exclusionary.
* Has body mass index (BMI) within the range of 18.5-31.0 kilograms per meter square (kg/m^2).
* Participants male at birth must use male condoms and participants female at birth who are of childbearing potential must be using acceptable forms of birth control.
* Participants capable of giving signed informed consent.
* Participant must be willing and able to start locally accessible and commercially available combination antiretroviral therapy after the monotherapy period.

Exclusion Criteria:

* Women who are breastfeeding or plan to become pregnant or breast feed during the study.
* Participants with acute HIV infection.
* Any evidence of an active Centers for Disease Control and Prevention (CDC) Stage 3 disease.
* Untreated syphilis infection.
* Ongoing malignancy other than certain localised malignancies.
* Treatment with immunomodulating agents or any agent with known anti-HIV activity.
* Has exclusionary psychiatric, hepatic, cardiovascular gastrointestinal, renal condition.
* Participant having any condition which, in the opinion of the investigator, may interfere with the absorption, distribution, metabolism or excretion of the study drugs or render the participant unable to take oral medication.
* Participants having exclusionary electrocardiogram (ECG) findings.
* Participants who have been exposed to any prohibited medication or vaccine.
* Participant positive for hepatitis B or hepatitis C.
* Participants with exclusionary safety laboratory (e.g Grade 3 or greater abnormality).
* Participants who have positive results for illicit drug use, regular use of drugs of abuse and/or excessive alcohol use.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (3):
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Newark, New Jersey
- Argentina (2):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Bueno
- GSK Investigational Site, Montreal, Quebec, Canada
- France (3):
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
- GSK Investigational Site, Cologne, Germany
- GSK Investigational Site, Milan, Italy
- Mexico (2):
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Mexico City
- Spain (2):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to: https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants that were enrolled started the study.
Period: Monotherapy (Day 1-Day 11)
Arm/Group | Part 1a: VH4004280 Dose Level 1 | Part 1a: VH4004280 Dose Level 2 | Part 2a: VH4004280 Pre-specified Dose | Matching Placebo for VH4004280 | Part 1b: VH4011499 Dose Level 1 | Part 1b: VH4011499 Dose Level 2 | Part 2b: VH4011499 Pre-specified Dose | Matching Placebo for VH4011499
Started | 6 | 6 | 6 | 3 | 7 | 6 | 7 | 3
Completed | 6 | 6 | 6 | 3 | 7 | 6 | 7 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Follow-Up (Day 11-Day 39)
Arm/Group | Part 1a: VH4004280 Dose Level 1 | Part 1a: VH4004280 Dose Level 2 | Part 2a: VH4004280 Pre-specified Dose | Matching Placebo for VH4004280 | Part 1b: VH4011499 Dose Level 1 | Part 1b: VH4011499 Dose Level 2 | Part 2b: VH4011499 Pre-specified Dose | Matching Placebo for VH4011499
Started | 6 | 6 | 6 | 3 | 7 | 6 | 7 | 3
Completed | 6 | 6 | 6 | 3 | 7 | 6 | 7 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline measures are presented based on Exposed population, which included all participants that received a study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1a: VH4004280 Dose Level 1 | Part 1a: VH4004280 Dose Level 2 | Part 2a: VH4004280 Pre-specified Dose | Matching Placebo for VH4004280 | Part 1b: VH4011499 Dose Level 1 | Part 1b: VH4011499 Dose Level 2 | Part 2b: VH4011499 Pre-specified Dose | Matching Placebo for VH4011499 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 7 | 6 | 7 | 3 | 44
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 34.3 (12.82) | 42.8 (10.3) | 31.5 (9.75) | 28.7 (9.29) | 31.6 (9.29) | 49.3 (7.45) | 28.6 (9.93) | 26 (2.65) | 34.8 (11.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 5 | 5 | 6 | 2 | 7 | 3 | 6 | 3 | 37
  Female | 1 | 1 | 0 | 1 | 0 | 3 | 1 | 0 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 4
  Black or African American | 1 | 2 | 2 | 0 | 0 | 3 | 0 | 1 | 9
  White | 5 | 4 | 4 | 3 | 7 | 3 | 3 | 2 | 31

OUTCOME MEASURES:

1. Primary Outcome: Monotherapy, VH4004280: Maximum Change From Baseline (Day 1) in Plasma HIV-1 Ribonucleic Acid (RNA) log10
Description: Plasma samples were collected for quantitative analysis of plasma HIV-1 RNA. Maximum change from baseline was calculated by subtracting the baseline value from the post-dose visit value when the plasma HIV-1 RNA reached its minimum level up to Day 11 (inclusive). Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. The results were expressed as log10 copies per milliliter (log10 c/mL).
Time Frame: From Baseline (Day 1) and up to Day 11
Population: Analysis was performed on Full Analysis Set (FAS) population, which included all randomized participants who received at least one full dose of study treatment. Only participants that received VH4004280 intervention or matching placebo for VH4004280 and had data available at the specified timepoints were included in this analysis.
Measure: Mean (Standard Deviation); unit: log10 c/mL
Arm/Group | Part 1a: VH4004280 Dose Level 1 | Part 1a: VH4004280 Dose Level 2 | Part 2a: VH4004280 Pre-specified Dose | Matching Placebo for VH4004280
Number analyzed (Participants) | 6 | 6 | 6 | 3
log10 c/mL
  Baseline (Day 1) | 5.004 (0.4592) | 4.923 (0.5428) | 4.866 (0.7696) | 4.636 (0.6641)
  Maximum change compared to Baseline (Day 1) | -1.056 (0.4567) | -1.391 (0.6986) | -1.983 (0.2171) | -0.070 (0.0574)

2. Primary Outcome: Monotherapy, VH4011499: Maximum Change From Baseline (Day 1) in Plasma HIV-1 RNA log10
Description: Plasma samples were collected for quantitative analysis of plasma HIV-1 RNA. Maximum change from baseline was calculated by subtracting the baseline value from the post-dose visit value when the plasma HIV-1 RNA reached its minimum level up to Day 11 (inclusive). Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: From Baseline (Day 1) and up to Day 11
Population: Analysis was performed on FAS population. Only participants that received VH4011499 intervention or matching placebo for VH4011499 and had data available at the specified timepoints were included in this analysis.
Measure: Mean (Standard Deviation); unit: log10 c/mL
Arm/Group | Part 1b: VH4011499 Dose Level 1 | Part 1b: VH4011499 Dose Level 2 | Part 2b: VH4011499 Pre-specified Dose | Matching Placebo for VH4011499
Number analyzed (Participants) | 7 | 6 | 7 | 3
log10 c/mL
  Baseline (Day 1) | 5.001 (0.7304) | 4.339 (0.6185) | 4.960 (0.7288) | 4.714 (0.7736)
  Maximum change compared to Baseline (Day 1) | -1.834 (0.5141) | -1.797 (0.4544) | -2.165 (0.4310) | -0.176 (0.1969)

3. Secondary Outcome: Monotherapy: Number of Participants With Any Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Any = occurrence of the event regardless of intensity grade or relation to the study intervention.
Time Frame: From Baseline (Day 1) and up to Day 11
Population: Analysis was performed on Safety Population, which included all randomized participants who received at least 1 dose of study treatment and had safety data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a: VH4004280 Dose Level 1 | Part 1a: VH4004280 Dose Level 2 | Part 2a: VH4004280 Pre-specified Dose | Matching Placebo for VH4004280 | Part 1b: VH4011499 Dose Level 1 | Part 1b: VH4011499 Dose Level 2 | Part 2b: VH4011499 Pre-specified Dose | Matching Placebo for VH4011499
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 7 | 6 | 7 | 3
Participants | 3 | 2 | 2 | 2 | 2 | 4 | 2 | 1

4. Secondary Outcome: Follow-up: Number of Participants With Any AEs
Description: as for outcome 3
Time Frame: From Day 11 and up to Day 39
Population: Analysis was performed on Safety Population.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1a: VH4004280 Dose Level 1: Participants received a single dose of VH4004280 Dose Level 1 (low concentration) on Day 1 (evaluated for a 10-day period). On Day 11, participants switched to an open-label ART up to day 39.
- Part 1b: VH4011499 Dose Level 1: Participants received a single dose of VH4011499 Dose Level 1 (low concentration) on Day 1 and Day 6 (evaluated for a 10-day period). On Day 11, participants switched to an open-label ART up to day 39.
Arm/Group | Part 1a: VH4004280 Dose Level 1 | Part 1a: VH4004280 Dose Level 2 | Part 2a: VH4004280 Pre-specified Dose | Matching Placebo for VH4004280 | Part 1b: VH4011499 Dose Level 1 | Part 1b: VH4011499 Dose Level 2 | Part 2b: VH4011499 Pre-specified Dose | Matching Placebo for VH4011499
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 7 | 6 | 7 | 3
Participants | 1 | 3 | 4 | 1 | 3 | 3 | 5 | 0

5. Secondary Outcome: Monotherapy: Number of Participants With AEs by Severity
Description: Severity was rated according to the Division of Acquired Immunodeficiency Syndrome (DAIDS) grading criteria, where Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = potentially life-threatening, Grade 5 = death.
Time Frame: From Baseline (Day 1) and up to Day 11
Population: Analysis was performed on Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a: VH4004280 Dose Level 1 | Part 1a: VH4004280 Dose Level 2 | Part 2a: VH4004280 Pre-specified Dose | Matching Placebo for VH4004280 | Part 1b: VH4011499 Dose Level 1 | Part 1b: VH4011499 Dose Level 2 | Part 2b: VH4011499 Pre-specified Dose | Matching Placebo for VH4011499
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 7 | 6 | 7 | 3
Participants
  Grade 1 | 0 | 2 | 1 | 1 | 1 | 3 | 2 | 1
  Grade 2 | 3 | 0 | 1 | 1 | 1 | 1 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Follow-up: Number of Participants With AEs by Severity
Description: Severity was rated according to the DAIDS grading criteria, where Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = potentially life-threatening, Grade 5 = death.
Time Frame: From Day 11 and up to Day 39
Population: Analysis was performed on Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a: VH4004280 Dose Level 1 | Part 1a: VH4004280 Dose Level 2 | Part 2a: VH4004280 Pre-specified Dose | Matching Placebo for VH4004280 | Part 1b: VH4011499 Dose Level 1 | Part 1b: VH4011499 Dose Level 2 | Part 2b: VH4011499 Pre-specified Dose | Matching Placebo for VH4011499
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 7 | 6 | 7 | 3
Participants
  Grade 1 | 1 | 1 | 1 | 0 | 2 | 1 | 2 | 0
  Grade 2 | 0 | 1 | 3 | 1 | 1 | 2 | 3 | 0
  Grade 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Monotherapy: Number of Participants With AEs Leading to Study Treatment Discontinuation
Description: 'Discontinuation' of study intervention refers to any participant who has not received all planned doses of study intervention.
Time Frame: From Baseline (Day 1) and up to Day 11
Population: Analysis was performed on Safety Population, which included all participants that received at least one study intervention. Discontinuation of treatment was not possible for participants that received VH4004280 or matching placebo for VH4004280, since these participants received only one dose intervention at Day 1 (all planned interventions as per protocol schedule).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a: VH4004280 Dose Level 1 | Part 1a: VH4004280 Dose Level 2 | Part 2a: VH4004280 Pre-specified Dose | Matching Placebo for VH4004280 | Part 1b: VH4011499 Dose Level 1 | Part 1b: VH4011499 Dose Level 2 | Part 2b: VH4011499 Pre-specified Dose | Matching Placebo for VH4011499
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 6 | 7 | 3
Participants |  |  |  |  | 0 | 0 | 0 | 0

8. Secondary Outcome: Monotherapy and Follow-up, VH4004280: Change From Baseline for Liver Panel Laboratory Parameters - Total Bilirubin and Direct Bilirubin
Description: Change from Baseline values for liver panel laboratory parameters total bilirubin and direct bilirubin were summarised. Change from baseline was calculated by subtracting the baseline value from the post-dose visit value.Standard deviation (SD) = 0.0000 is defined as following: if all participants analyzed for a specific parameter at a specific time point have the same value, then SD is equal with 0.0000.
Time Frame: At Baseline (Day 1) and at Days 2, 4, 6, 7, 9, 11, 18, 25, 32 and 39
Population: Analysis was performed on Safety Population. Only participants that received VH4004280 intervention or matching placebo for VH4004280 and had data available at the specified timepoints were included in the analysis.
Measure: Mean (Standard Deviation); unit: Micromole per liter (µmol/L)
Arm/Group | Part 1a: VH4004280 Dose Level 1 | Part 1a: VH4004280 Dose Level 2 | Part 2a: VH4004280 Pre-specified Dose | Matching Placebo for VH4004280
Number analyzed (Participants) | 6 | 6 | 6 | 3
Micromole per liter (µmol/L)
  Total Bilirubin, Baseline (Day 1) | 6.641 (1.5157) | 8.408 (5.5383) | 6.926 (4.6300) | 6.783 (1.2370)
  Total Bilirubin, Day 2: number analyzed (Participants) | 6 | 6 | 5 | 3
  Total Bilirubin, Day 2 | -0.143 (1.7719) | -0.513 (2.9697) | 0.239 (4.4814) | 1.995 (3.5100)
  Total Bilirubin, Day 4: number analyzed (Participants) | 5 | 6 | 5 | 3
  Total Bilirubin, Day 4 | 0.547 (1.0073) | -2.081 (3.5614) | 1.984 (3.1078) | -1.767 (1.5516)
  Total Bilirubin, Day 6 | -0.171 (3.5771) | 0.485 (3.6055) | 2.366 (5.2755) | 2.565 (2.8460)
  Total Bilirubin, Day 7 | 1.539 (1.4307) | 0.941 (3.3295) | 0.599 (2.4774) | 1.767 (3.2189)
  Total Bilirubin, Day 9: number analyzed (Participants) | 5 | 6 | 6 | 3
  Total Bilirubin, Day 9 | 1.060 (2.5230) | 0.656 (4.2584) | 1.055 (1.7752) | 0.969 (3.7672)
  Total Bilirubin, Day 11: number analyzed (Participants) | 4 | 6 | 6 | 3
  Total Bilirubin, Day 11 | 1.154 (1.5758) | 1.539 (1.8670) | 0.085 (1.2649) | -0.171 (2.7360)
  Total Bilirubin, Day 18 | 0.684 (2.6513) | 0.399 (2.4005) | -1.340 (3.2199) | -0.342 (1.8016)
  Total Bilirubin, Day 25 | 0.570 (1.1731) | 0.513 (3.0049) | -2.195 (3.5417) | -0.741 (2.2771)
  Total Bilirubin, Day 32 | 0.770 (2.1596) | -0.542 (2.5557) | -1.881 (3.4709) | 1.026 (3.6194)
  Total Bilirubin, Day 39: number analyzed (Participants) | 5 | 6 | 5 | 3
  Total Bilirubin, Day 39 | 0.923 (1.3712) | -1.197 (3.2910) | -0.513 (3.2332) | 0.456 (2.8682)
  Direct Bilirubin, Baseline (Day 1) | 3.410 (0.0000) | 3.410 (0.0000) | 3.410 (0.0000) | 3.410 (0.0000)
  Direct Bilirubin, Day 2 | 0.000 (0.0000) | 0.002 (0.0041) | 0.000 (0.0000) | 0.000 (0.0000)
  Direct Bilirubin, Day 4: number analyzed (Participants) | 5 | 6 | 6 | 3
  Direct Bilirubin, Day 4 | 0.000 (0.0000) | 0.000 (0.0000) | 0.002 (0.0041) | 0.000 (0.0000)
  Direct Bilirubin, Day 6 | 0.000 (0.0000) | 0.030 (0.0739) | 0.030 (0.0739) | 0.000 (0.0000)
  Direct Bilirubin, Day 7 | 0.000 (0.0000) | 0.059 (0.1437) | 0.000 (0.0000) | 0.000 (0.0000)
  Direct Bilirubin, Day 9: number analyzed (Participants) | 5 | 6 | 6 | 3
  Direct Bilirubin, Day 9 | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Direct Bilirubin, Day 11: number analyzed (Participants) | 4 | 6 | 6 | 3
  Direct Bilirubin, Day 11 | 0.000 (0.0000) | 0.002 (0.0041) | 0.000 (0.0000) | 0.000 (0.0000)
  Direct Bilirubin, Day 18: number analyzed (Participants) | 6 | 6 | 5 | 3
  Direct Bilirubin, Day 18 | 0.000 (0.0000) | 0.174 (0.4221) | 0.000 (0.0000) | 0.000 (0.0000)
  Direct Bilirubin, Day 25 | 0.000 (0.0000) | 0.030 (0.0739) | 0.000 (0.0000) | 0.000 (0.0000)
  Direct Bilirubin, Day 32: number analyzed (Participants) | 5 | 5 | 6 | 3
  Direct Bilirubin, Day 32 | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Direct Bilirubin, Day 39: number analyzed (Participants) | 5 | 6 | 6 | 3
  Direct Bilirubin, Day 39 | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)

9. Secondary Outcome: Monotherapy and Follow-up, VH4011499: Change From Baseline for Liver Panel Laboratory Parameters - Total Bilirubin and Direct Bilirubin
Description: Change from Baseline values for liver panel laboratory parameters total bilirubin and direct bilirubin were summarised. Change from baseline was calculated by subtracting the baseline value from the post-dose visit value. SD = 0.0000 is defined as following: if all participants analyzed for a specific parameter at a specific time point have the same value, then SD is equal with 0.0000.
Time Frame: At Baseline (Day 1) and at Days 2, 4, 6, 7, 9, 11, 18, 25, 32 and 39
Population: Analysis was performed on Safety Population. Only participants that received VH4011499 intervention or matching placebo for VH4011499 and had data available at the specified timepoints were included in the analysis.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Part 1b: VH4011499 Dose Level 1 | Part 1b: VH4011499 Dose Level 2 | Part 2b: VH4011499 Pre-specified Dose | Matching Placebo for VH4011499
Number analyzed (Participants) | 7 | 6 | 7 | 3
µmol/L
  Total Bilirubin, Baseline (Day 1) | 5.643 (2.4898) | 7.524 (2.6579) | 4.544 (1.7576) | 7.011 (2.2361)
  Total Bilirubin, Day 2 | -0.928 (0.9095) | 0.114 (0.9951) | 0.611 (1.6008) | -0.855 (0.6165)
  Total Bilirubin, Day 4 | 0.122 (2.3975) | -0.656 (0.9937) | 1.808 (2.3463) | -0.570 (1.5516)
  Total Bilirubin, Day 6 | -0.171 (2.4741) | -1.967 (2.6286) | 0.440 (1.4370) | -2.109 (3.6529)
  Total Bilirubin, Day 7 | 0.366 (3.4476) | -0.200 (2.7111) | 0.367 (1.4081) | -1.995 (3.6569)
  Total Bilirubin, Day 9 | -0.440 (2.3774) | -0.228 (1.4004) | 1.099 (1.4804) | 0.912 (3.5924)
  Total Bilirubin, Day 11 | 1.050 (2.0766) | -0.884 (1.3439) | 0.709 (2.3036) | -2.964 (1.2370)
  Total Bilirubin, Day 18 | -0.366 (2.7081) | -0.057 (1.7989) | 0.586 (1.7739) | 1.083 (3.4427)
  Total Bilirubin, Day 25 | 0.366 (3.9024) | 0.798 (3.2258) | 1.295 (2.1332) | -1.026 (3.0059)
  Total Bilirubin, Day 32: number analyzed (Participants) | 6 | 6 | 7 | 3
  Total Bilirubin, Day 32 | 0.599 (2.9175) | 0.513 (3.3017) | 1.075 (2.2398) | 0.627 (4.9452)
  Total Bilirubin, Day 39: number analyzed (Participants) | 5 | 6 | 7 | 2
  Total Bilirubin, Day 39 | 0.239 (1.3927) | -0.599 (1.7861) | 0.489 (2.2630) | -0.855 (0.2418)
  Direct Bilirubin, Baseline (Day 1) | 3.485 (0.1977) | 3.410 (0.0000) | 3.705 (0.7794) | 3.527 (0.2032)
  Direct Bilirubin, Day 2 | -0.075 (0.1977) | 0.000 (0.0000) | -0.295 (0.7794) | -0.117 (0.2032)
  Direct Bilirubin, Day 4: number analyzed (Participants) | 6 | 6 | 7 | 3
  Direct Bilirubin, Day 4 | -0.057 (0.1396) | 0.000 (0.0000) | -0.295 (0.7794) | -0.114 (0.1975)
  Direct Bilirubin, Day 6 | -0.073 (0.1939) | 0.000 (0.0000) | -0.295 (0.7794) | -0.117 (0.2032)
  Direct Bilirubin, Day 7 | -0.049 (0.2197) | 0.000 (0.0000) | -0.295 (0.7794) | 1.140 (2.2862)
  Direct Bilirubin, Day 9 | -0.075 (0.1977) | 0.002 (0.0041) | -0.295 (0.7794) | -0.057 (0.0987)
  Direct Bilirubin, Day 11 | -0.073 (0.1983) | 0.000 (0.0000) | -0.295 (0.7794) | -0.117 (0.2032)
  Direct Bilirubin, Day 18 | -0.075 (0.1977) | 0.000 (0.0000) | -0.295 (0.7794) | 0.057 (0.0987)
  Direct Bilirubin, Day 25 | 0.027 (0.1571) | 0.030 (0.0739) | -0.295 (0.7794) | -0.114 (0.1975)
  Direct Bilirubin, Day 32: number analyzed (Participants) | 6 | 6 | 7 | 3
  Direct Bilirubin, Day 32 | -0.057 (0.2395) | 0.230 (0.5626) | -0.295 (0.7794) | 0.114 (0.1975)
  Direct Bilirubin, Day 39: number analyzed (Participants) | 6 | 6 | 7 | 2
  Direct Bilirubin, Day 39 | -0.087 (0.2135) | 0.000 (0.0000) | -0.295 (0.7794) | -0.171 (0.2418)

10. Secondary Outcome: Monotherapy and Follow-up, VH4004280: Change From Baseline for Liver Panel Laboratory Parameters - Alanine Aminotransferace (ALT), Alkaline Phosphatase (ALP) and Aspartate Aminotransferase (AST)
Description: Change from Baseline values for liver panel laboratory parameters ALT, ALP and AST were summarised. Change from baseline was calculated by subtracting the baseline value from the post-dose visit value.
Time Frame: At Baseline (Day 1) and at Days 2, 4, 6, 7, 9, 11, 18, 25, 32 and 39
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Part 1a: VH4004280 Dose Level 1 | Part 1a: VH4004280 Dose Level 2 | Part 2a: VH4004280 Pre-specified Dose | Matching Placebo for VH4004280
Number analyzed (Participants) | 6 | 6 | 6 | 3
International units per liter (IU/L)
  ALT, Baseline (Day 1) | 31.3 (13.59) | 21.7 (7.17) | 33.2 (13.23) | 52.7 (55.82)
  ALT, Day 2: number analyzed (Participants) | 6 | 6 | 5 | 3
  ALT, Day 2 | -2.8 (3.25) | -1.8 (3.25) | -0.2 (3.56) | 15.0 (29.46)
  ALT, Day 4: number analyzed (Participants) | 5 | 6 | 5 | 3
  ALT, Day 4 | -3.8 (4.09) | -2.3 (2.80) | 0.2 (6.10) | 4.7 (9.29)
  ALT, Day 6 | -7.8 (9.33) | -1.3 (1.51) | 2.2 (8.13) | -13.7 (27.14)
  ALT, Day 7 | -6.7 (9.77) | -2.0 (3.03) | 0.2 (7.39) | -19.3 (32.62)
  ALT, Day 9: number analyzed (Participants) | 5 | 6 | 6 | 3
  ALT, Day 9 | -6.0 (13.69) | -0.7 (9.63) | 1.5 (12.10) | -20.7 (35.81)
  ALT, Day 11: number analyzed (Participants) | 4 | 6 | 6 | 3
  ALT, Day 11 | -8.8 (15.78) | -2.0 (6.26) | -0.2 (11.99) | -16.7 (29.74)
  ALT, Day 18 | -6.2 (14.16) | -0.2 (4.45) | 8.3 (27.46) | -15.7 (31.18)
  ALT, Day 25 | -6.8 (15.48) | -0.5 (2.17) | 1.7 (14.54) | -27.7 (44.50)
  ALT, Day 32 | -9.2 (11.97) | -0.3 (4.23) | 0.3 (12.32) | -33.0 (56.40)
  ALT, Day 39: number analyzed (Participants) | 5 | 6 | 5 | 3
  ALT, Day 39 | -9.8 (11.12) | -0.3 (3.50) | -4.0 (8.72) | -33.0 (54.62)
  ALP, Baseline (Day 1) | 79.2 (14.40) | 74.3 (15.74) | 71.7 (19.39) | 64.3 (16.80)
  ALP, Day 2: number analyzed (Participants) | 6 | 6 | 5 | 3
  ALP, Day 2 | -1.3 (7.87) | -2.7 (10.03) | -1.0 (3.16) | -3.0 (3.00)
  ALP, Day 4: number analyzed (Participants) | 5 | 6 | 5 | 3
  ALP, Day 4 | 0.6 (5.41) | -5.0 (5.90) | -2.6 (2.51) | -1.0 (3.61)
  ALP, Day 6 | 1.5 (6.75) | -4.5 (6.35) | 0.7 (5.35) | -2.3 (1.15)
  ALP, Day 7 | -0.2 (6.24) | -6.2 (2.71) | -2.0 (4.52) | -6.0 (4.36)
  ALP, Day 9: number analyzed (Participants) | 5 | 6 | 6 | 3
  ALP, Day 9 | -0.2 (2.95) | -4.3 (6.09) | -3.5 (5.82) | -6.3 (6.66)
  ALP, Day 11: number analyzed (Participants) | 4 | 6 | 6 | 3
  ALP, Day 11 | -5.0 (2.94) | -4.8 (6.05) | -5.8 (8.28) | -6.3 (4.93)
  ALP, Day 18 | -0.5 (3.33) | -7.0 (5.40) | -2.7 (8.50) | -4.3 (4.51)
  ALP, Day 25 | 1.0 (11.17) | -5.0 (4.69) | -1.3 (8.71) | -5.0 (4.36)
  ALP, Day 32 | 3.2 (21.10) | -2.7 (10.84) | -3.8 (8.47) | -5.3 (5.77)
  ALP, Day 39: number analyzed (Participants) | 5 | 6 | 5 | 3
  ALP, Day 39 | 0.6 (4.16) | -5.5 (7.82) | -2.2 (4.15) | 0.3 (3.51)
  AST, Baseline (Day 1) | 26.0 (4.94) | 21.5 (4.23) | 27.2 (3.49) | 29.7 (11.72)
  AST, Day 2: number analyzed (Participants) | 6 | 6 | 5 | 3
  AST, Day 2 | -3.5 (3.62) | -0.8 (2.71) | -0.2 (4.09) | 11.0 (26.00)
  AST, Day 4: number analyzed (Participants) | 5 | 6 | 5 | 3
  AST, Day 4 | -3.6 (3.21) | -0.8 (0.75) | 0.8 (3.96) | -1.0 (5.29)
  AST, Day 6 | -4.8 (4.36) | -2.0 (1.26) | 0.7 (5.54) | -8.3 (11.06)
  AST, Day 7 | -4.8 (4.54) | -2.2 (2.23) | -1.2 (4.88) | -9.0 (9.85)
  AST, Day 9: number analyzed (Participants) | 5 | 6 | 6 | 3
  AST, Day 9 | -5.0 (6.00) | -1.5 (4.72) | 2.5 (8.53) | -9.3 (10.69)
  AST, Day 11: number analyzed (Participants) | 4 | 6 | 6 | 3
  AST, Day 11 | -6.3 (6.34) | -2.0 (4.60) | 7.0 (22.52) | -6.7 (5.03)
  AST, Day 18 | -4.7 (6.44) | 0.0 (6.51) | 4.2 (16.46) | -1.0 (3.61)
  AST, Day 25 | -4.7 (9.35) | -0.3 (3.56) | 1.5 (7.40) | -11.3 (11.93)
  AST, Day 32 | -5.0 (6.81) | -1.3 (3.08) | 0.7 (4.72) | -9.0 (14.80)
  AST, Day 39: number analyzed (Participants) | 5 | 6 | 5 | 3
  AST, Day 39 | -6.6 (5.50) | 0.5 (3.39) | -2.4 (3.13) | -10.3 (13.65)

11. Secondary Outcome: Monotherapy and Follow-up, VH4011499: Change From Baseline for Liver Panel Laboratory Parameters - ALT, ALP and AST
Description: as for outcome 10
Time Frame: At Baseline (Day 1) and at Days 2, 4, 6, 7, 9, 11, 18, 25, 32 and 39
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Part 1b: VH4011499 Dose Level 1 | Part 1b: VH4011499 Dose Level 2 | Part 2b: VH4011499 Pre-specified Dose | Matching Placebo for VH4011499
Number analyzed (Participants) | 7 | 6 | 7 | 3
IU/L
  ALT, Baseline (Day 1) | 14.9 (4.41) | 19.5 (9.03) | 31.7 (22.60) | 18.3 (2.08)
  ALT, Day 2 | 1.7 (1.25) | -1.2 (1.83) | -1.6 (3.78) | 0.7 (0.58)
  ALT, Day 4 | 2.4 (1.72) | -1.0 (3.85) | -3.6 (13.20) | -1.0 (1.00)
  ALT, Day 6 | -0.1 (1.57) | -1.2 (3.76) | -5.1 (14.58) | 0.7 (1.15)
  ALT, Day 7 | 0.1 (2.54) | -1.5 (4.76) | -7.3 (14.91) | -0.7 (1.57)
  ALT, Day 9 | -0.3 (1.98) | -0.2 (4.07) | -8.0 (16.42) | -0.3 (2.08)
  ALT, Day 11 | 0.0 (3.32) | -1.2 (3.76) | -7.3 (11.71) | 0.0 (3.61)
  ALT, Day 18 | 0.3 (5.19) | -1.3 (4.46) | -4.0 (17.91) | 1.7 (2.52)
  ALT, Day 25 | 2.0 (9.02) | 0.0 (5.66) | -7.4 (17.52) | 0.7 (0.58)
  ALT, Day 32: number analyzed (Participants) | 6 | 6 | 7 | 3
  ALT, Day 32 | 4.0 (13.62) | -2.7 (3.88) | -10.3 (16.63) | 3.0 (4.36)
  ALT, Day 39: number analyzed (Participants) | 5 | 6 | 7 | 2
  ALT, Day 39 | 0.0 (7.84) | 0.8 (4.49) | -3.6 (15.87) | 28.0 (28.28)
  ALP, Baseline (Day 1) | 81.1 (14.55) | 68.2 (18.90) | 78.9 (20.69) | 89.3 (16.50)
  ALP, Day 2 | 1.0 (5.60) | -1.2 (2.48) | 0.6 (6.48) | -0.3 (1.53)
  ALP, Day 4 | 2.7 (6.97) | -2.5 (3.33) | -4.9 (13.38) | -0.7 (7.51)
  ALP, Day 6 | -1.4 (7.44) | -3.7 (5.75) | -3.6 (4.69) | 6.3 (8.33)
  ALP, Day 7 | 3.9 (5.70) | -4.5 (3.39) | -0.4 (8.66) | 4.0 (8.72)
  ALP, Day 9 | 0.0 (9.80) | -1.5 (1.76) | -1.4 (9.76) | -0.7 (8.08)
  ALP, Day 11 | 2.9 (13.32) | -1.3 (3.20) | -1.6 (7.96) | 10.3 (14.47)
  ALP, Day 18 | -0.1 (6.01) | -3.2 (3.92) | -2.9 (6.49) | 2.3 (9.71)
  ALP, Day 25 | 2.4 (7.59) | -5.0 (5.76) | -6.4 (10.97) | -1.7 (17.21)
  ALP, Day 32: number analyzed (Participants) | 6 | 6 | 7 | 3
  ALP, Day 32 | 0.3 (9.05) | -4.5 (3.45) | -3.7 (9.81) | -2.3 (8.02)
  ALP, Day 39: number analyzed (Participants) | 5 | 6 | 7 | 2
  ALP, Day 39 | -2.4 (13.72) | -2.2 (8.04) | -1.7 (14.69) | 1.0 (11.31)
  AST, Baseline (Day 1) | 18.6 (3.87) | 24.0 (8.07) | 24.7 (7.20) | 27.7 (5.51)
  AST, Day 2 | -0.7 (2.43) | -2.3 (2.80) | -2.0 (1.29) | -2.3 (3.21)
  AST, Day 4 | 1.1 (4.45) | -2.7 (3.27) | 1.7 (7.50) | -2.3 (0.58)
  AST, Day 6 | -0.9 (4.02) | -1.5 (5.68) | -2.4 (3.55) | -1.7 (3.21)
  AST, Day 7 | -1.7 (4.07) | -3.5 (5.75) | -3.7 (5.12) | -5.7 (2.31)
  AST, Day 9 | 0.0 (3.00) | -2.7 (4.41) | -4.3 (5.02) | -5.0 (6.24)
  AST, Day 11 | -1.6 (3.74) | -2.2 (4.79) | -2.1 (3.29) | -4.7 (7.51)
  AST, Day 18 | -1.3 (5.82) | -3.2 (5.31) | 2.4 (9.55) | -0.3 (5.51)
  AST, Day 25 | 1.6 (5.86) | -0.5 (4.32) | -2.6 (4.86) | -3.7 (0.58)
  AST, Day 32: number analyzed (Participants) | 6 | 5 | 7 | 3
  AST, Day 32 | 2.8 (9.97) | -1.4 (3.13) | -2.9 (6.69) | -2.3 (4.93)
  AST, Day 39: number analyzed (Participants) | 5 | 6 | 7 | 2
  AST, Day 39 | 0.0 (5.43) | 1.3 (2.58) | 1.7 (10.64) | 23.0 (5.66)

12. Secondary Outcome: Monotherapy and Follow-up, VH4004280: Number of Participants With Maximum Toxicity Grade Increase From Baseline for Liver Panel Laboratory Parameters - Total Bilirubin and Direct Bilirubin
Description: Laboratory abnormalities were graded according to DAIDS grading table Version 2.1 where grades were defined based on numeric criteria as follows Grade 0: participants with missing baseline values; Grade 1: Mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences.
Time Frame: From Baseline (Day 1) and up to Day 39
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a: VH4004280 Dose Level 1 | Part 1a: VH4004280 Dose Level 2 | Part 2a: VH4004280 Pre-specified Dose | Matching Placebo for VH4004280
Number analyzed (Participants) | 6 | 6 | 6 | 3
Participants
  Total Bilirubin, Increase to Grade 1 | 0 | 1 | 0 | 0
  Total Bilirubin, Increase to Grade 2 | 0 | 0 | 0 | 0
  Total Bilirubin, Increase to Grade 3 | 0 | 0 | 0 | 0
  Total Bilirubin, Increase to Grade 4 | 0 | 0 | 0 | 0
  Direct Bilirubin, Increase to Grade 1 | 0 | 0 | 0 | 0
  Direct Bilirubin, Increase to Grade 2 | 0 | 0 | 0 | 0
  Direct Bilirubin, Increase to Grade 3 | 0 | 0 | 0 | 0
  Direct Bilirubin, Increase to Grade 4 | 0 | 0 | 0 | 0

13. Secondary Outcome: Monotherapy and Follow-up, VH4011499: Number of Participants With Maximum Toxicity Grade Increase From Baseline for Liver Panel Laboratory Parameters - Total Bilirubin and Direct Bilirubin
Description: as for outcome 12
Time Frame: From Baseline (Day 1) and up to Day 39
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1b: VH4011499 Dose Level 1 | Part 1b: VH4011499 Dose Level 2 | Part 2b: VH4011499 Pre-specified Dose | Matching Placebo for VH4011499
Number analyzed (Participants) | 7 | 6 | 7 | 3
Participants
  Total Bilirubin, Increase to Grade 1 | 0 | 0 | 0 | 0
  Total Bilirubin, Increase to Grade 2 | 0 | 0 | 0 | 0
  Total Bilirubin, Increase to Grade 3 | 0 | 0 | 0 | 0
  Total Bilirubin, Increase to Grade 4 | 0 | 0 | 0 | 0
  Direct Bilirubin, Increase to Grade 1 | 0 | 0 | 0 | 0
  Direct Bilirubin, Increase to Grade 2 | 0 | 0 | 0 | 0
  Direct Bilirubin, Increase to Grade 3 | 0 | 0 | 0 | 1
  Direct Bilirubin, Increase to Grade 4 | 0 | 0 | 0 | 0

14. Secondary Outcome: Monotherapy and Follow-up, VH4004280: Number of Participants With Maximum Toxicity Grade Increase From Baseline for Liver Panel Laboratory Parameters - ALT, ALP and AST
Description: as for outcome 12
Time Frame: From Baseline (Day 1) and up to Day 39
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a: VH4004280 Dose Level 1 | Part 1a: VH4004280 Dose Level 2 | Part 2a: VH4004280 Pre-specified Dose | Matching Placebo for VH4004280
Number analyzed (Participants) | 6 | 6 | 6 | 3
Participants
  ALT, Increase to Grade 1 | 1 | 0 | 1 | 0
  ALT, Increase to Grade 2 | 0 | 0 | 1 | 0
  ALT, Increase to Grade 3 | 0 | 0 | 0 | 0
  ALT, Increase to Grade 4 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 1 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 2 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 3 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 4 | 0 | 0 | 0 | 0
  AST, Increase to Grade 1 | 1 | 0 | 1 | 1
  AST, Increase to Grade 2 | 0 | 0 | 0 | 0
  AST, Increase to Grade 3 | 0 | 0 | 0 | 0
  AST, Increase to Grade 4 | 0 | 0 | 0 | 0

15. Secondary Outcome: Monotherapy and Follow-up, VH4011499: Number of Participants With Maximum Toxicity Grade Increase From Baseline for Liver Panel Laboratory Parameters - ALT, ALP and AST
Description: as for outcome 12
Time Frame: From Baseline (Day 1) and up to Day 39
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1b: VH4011499 Dose Level 1 | Part 1b: VH4011499 Dose Level 2 | Part 2b: VH4011499 Pre-specified Dose | Matching Placebo for VH4011499
Number analyzed (Participants) | 7 | 6 | 7 | 3
Participants
  ALT, Increase to Grade 1 | 0 | 0 | 1 | 1
  ALT, Increase to Grade 2 | 0 | 0 | 0 | 0
  ALT, Increase to Grade 3 | 0 | 0 | 0 | 0
  ALT, Increase to Grade 4 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 1 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 2 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 3 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 4 | 0 | 0 | 0 | 0
  AST, Increase to Grade 1 | 0 | 0 | 0 | 1
  AST, Increase to Grade 2 | 0 | 0 | 0 | 0
  AST, Increase to Grade 3 | 0 | 0 | 0 | 0
  AST, Increase to Grade 4 | 0 | 0 | 0 | 0

16. Secondary Outcome: Monotherapy, VH4004280: Maximum Observed Plasma Drug Concentration (Cmax)
Description: Cmax is defined as the maximum concentration of the drug in plasma.
Time Frame: After dose administration at Day 1
Population: Analysis was performed on Pharmacokinetic (PK) population, which included all participants in the Safety analysis population who had at least 1 non-missing PK assessment. Data was reported according to the actual study treatment. Only participants that received VH4004280 intervention and had data available at the specified timepoint were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Part 1a: VH4004280 Dose Level 1 | Part 1a: VH4004280 Dose Level 2 | Part 2a: VH4004280 Pre-specified Dose
Number analyzed (Participants) | 6 | 6 | 6
Nanogram per milliliter (ng/mL) | 131.57 (77.68) | 364.70 (85.21) | 473.00 (54.23)

17. Secondary Outcome: Monotherapy, VH4011499: Cmax
Description: Cmax is defined as the maximum concentration of the drug in plasma.
Time Frame: After dose administration at Day 1 and Day 6
Population: Analysis was performed on PK population. Only participants that received VH4011499 intervention and had data available at the specified timepoints were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1b: VH4011499 Dose Level 1 | Part 1b: VH4011499 Dose Level 2 | Part 2b: VH4011499 Pre-specified Dose
Number analyzed (Participants) | 7 | 6 | 7
ng/mL
  Day 1 | 27.63 (94.53) | 31.88 (26.58) | 133.59 (42.34)
  Day 6 | 35.30 (81.31) | 32.31 (25.97) | 141.18 (47.79)

18. Secondary Outcome: Monotherapy, VH4004280: Time to Maximum Observed Plasma Drug Concentration (Tmax)
Description: Tmax is a measure of the time required to reach the maximum concentration of the drug.
Time Frame: After dose administration at Day 1
Population: Analysis was performed on PK population. Only participants that received VH4004280 intervention and had data available at the specified timepoint were included in the analysis.
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Part 1a: VH4004280 Dose Level 1 | Part 1a: VH4004280 Dose Level 2 | Part 2a: VH4004280 Pre-specified Dose
Number analyzed (Participants) | 6 | 6 | 6
Hour (h) | 7.95 [6.0 to 9.7] | 9.00 [6.0 to 11.6] | 8.04 [6.0 to 10.0]

19. Secondary Outcome: Monotherapy, VH4011499: Tmax
Description: Tmax is a measure of the time required to reach the maximum concentration of the drug.
Time Frame: After dose administration at Day 1 and Day 6
Population: as for outcome 17
Measure: Median (Full Range); unit: h
Arm/Group | Part 1b: VH4011499 Dose Level 1 | Part 1b: VH4011499 Dose Level 2 | Part 2b: VH4011499 Pre-specified Dose
Number analyzed (Participants) | 7 | 6 | 7
h
  Day 1 | 9.95 [6.0 to 12.0] | 9.88 [8.1 to 10.1] | 8.00 [4.1 to 12.0]
  Day 6 | 10.00 [8.0 to 26.9] | 10.04 [8.0 to 11.6] | 11.52 [6.0 to 24.1]

20. Secondary Outcome: Monotherapy, VH4004280: Plasma Concentration at Day 11 (C11)
Description: C11 is defined as the concentration of the drug in plasma at Day 11.
Time Frame: At Day 11
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1a: VH4004280 Dose Level 1 | Part 1a: VH4004280 Dose Level 2 | Part 2a: VH4004280 Pre-specified Dose
Number analyzed (Participants) | 3 | 6 | 6
ng/mL | 18.07 (132.07) | 48.53 (130.33) | 50.42 (41.52)

21. Secondary Outcome: Monotherapy, VH4011499: C11
Description: C11 is defined as the concentration of the drug in plasma at Day 11.
Time Frame: At Day 11
Population: Analysis was performed on PK population. Only participants that received VH4011499 intervention and had data available at the specified timepoint were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1b: VH4011499 Dose Level 1 | Part 1b: VH4011499 Dose Level 2 | Part 2b: VH4011499 Pre-specified Dose
Number analyzed (Participants) | 6 | 4 | 7
ng/mL | 11.16 (50.02) | 10.56 (36.61) | 27.04 (50.68)

22. Secondary Outcome: Monotherapy, VH4004280: Change in Plasma HIV-1 RNA From Baseline
Description: Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from baseline was calculated by subtracting the baseline value from the post-dose visit value.
Time Frame: At Baseline (Day 1) and Day 11
Population: Analysis was performed on FAS population. Only participants that received VH4004280 intervention and had data available at the specified timepoints were included in the analysis.
Measure: Mean (Standard Deviation); unit: log10 c/mL
Arm/Group | Part 1a: VH4004280 Dose Level 1 | Part 1a: VH4004280 Dose Level 2 | Part 2a: VH4004280 Pre-specified Dose
Number analyzed (Participants) | 6 | 6 | 6
log10 c/mL
  Baseline (Day 1) | 5.004 (0.4592) | 4.923 (0.5428) | 4.866 (0.7696)
  Day 11: number analyzed (Participants) | 4 | 6 | 6
  Day 11 | -0.941 (0.6608) | -1.322 (0.7727) | -1.939 (0.1124)

23. Secondary Outcome: Monotherapy, VH4011499: Change in Plasma HIV-1 RNA From Baseline
Description: as for outcome 22
Time Frame: At Baseline (Day 1) and Day 11
Population: Analysis was performed on FAS population. Only participants that received VH4011499 intervention and had data available at the specified timepoints were included in the analysis.
Measure: Mean (Standard Deviation); unit: log10 c/mL
Arm/Group | Part 1b: VH4011499 Dose Level 1 | Part 1b: VH4011499 Dose Level 2 | Part 2b: VH4011499 Pre-specified Dose
Number analyzed (Participants) | 7 | 6 | 7
log10 c/mL
  Baseline (Day 1) | 5.001 (0.7304) | 4.339 (0.6185) | 4.960 (0.7288)
  Day 11 | -1.801 (0.5165) | -1.750 (0.4962) | -2.165 (0.4310)

ADVERSE EVENTS:
Time Frame: All-cause mortality, SAEs and non-serious AEs (including solicited and unsolicited events) were assessed from Day 1 [Monotherapy Phase] and up to Day 39 [Follow-up Phase].
Description: Adverse events are presented phase-wise (for Monotherapy and Follow-up phases), for the Exposed set, which included all participants that received at least one study dose administration.
Groups:
- Part 1a: VH4004280 Dose Level 1 (Monotherapy); Part 1a: VH4004280 Dose Level 1 (Follow-up): Participants received a single dose of VH4004280 Dose Level 1 (low concentration) on Day 1 (evaluated for a 10-day period). On Day 11, participants switched to an open-label antiretroviral therapy (ART) up to day 39.
- Part 2a: VH4004280 Pre-specified Dose (Monotherapy); Part 2a: VH4004280 Pre-specified Dose (Follow-up): Participants received a single pre-specified dose of VH4004280 (high concentration) on Day 1 (evaluated for a 10-day period). On Day 11, participants switched to an open-label ART up to day 39.
- Matching Placebo for VH4004280 (Monotherapy); Matching Placebo for VH4004280 (Follow-up): Participants received a matching placebo for VH4004280 on Day 1 (evaluated for a 10-day period). On Day 11, participants switched to an open-label ART up to day 39.
- Part 1b: VH4011499 Dose Level 1 (Monotherapy); Part 1b: VH4011499 Dose Level 1 (Follow-up): Participants received a single dose of VH4011499 Dose Level 1 (low concentration) on Day 1 and Day 6 (evaluated for a 10-day period). On Day 11, participants had the option to switch to an open-label ART up to day 39.
- Part 1b: VH4011499 Dose Level 2 (Monotherapy); Part 1b: VH4011499 Dose Level 2 (Follow-up): Participants received a single dose of VH4011499 Dose Level 2 (medium concentration) on Day 1 and Day 6 (evaluated for a 10-day period). On Day 11, participants switched to an open-label ART up to day 39.
- Part 2b: VH4011499 Pre-specified Dose (Monotherapy); Part 2b: VH4011499 Pre-specified Dose (Follow-up): Participants received a single pre-specified dose of VH4011499 (high concentration) on Day 1 and Day 6 (evaluated for a 10-day period). On Day 11, participants switched to an open-label ART up to day 39.
- Matching Placebo for VH4011499 (Monotherapy); Matching Placebo for VH4011499 (Follow-up): Participants received a matching placebo for VH4011499 on Day 1 and Day 6 (evaluated for a 10-day period). On Day 11, participants switched to an open-label ART up to day 39.
- Part 1a: VH4004280 Dose Level 2 (Follow-up): Participants received a single dose of VH4004280 Dose Level 2 (medium concentration) on Day 1 (evaluated for a 10-day period). On Day 11, participants switched to an open-label ART up to day 39.
Arm/Group | Part 1a: VH4004280 Dose Level 1 (Monotherapy) | Part 1a: VH4004280 Dose Level 2 | Part 2a: VH4004280 Pre-specified Dose (Monotherapy) | Matching Placebo for VH4004280 (Monotherapy) | Part 1b: VH4011499 Dose Level 1 (Monotherapy) | Part 1b: VH4011499 Dose Level 2 (Monotherapy) | Part 2b: VH4011499 Pre-specified Dose (Monotherapy) | Matching Placebo for VH4011499 (Monotherapy) | Part 1a: VH4004280 Dose Level 1 (Follow-up) | Part 1a: VH4004280 Dose Level 2 (Follow-up) | Part 2a: VH4004280 Pre-specified Dose (Follow-up) | Matching Placebo for VH4004280 (Follow-up) | Part 1b: VH4011499 Dose Level 1 (Follow-up) | Part 1b: VH4011499 Dose Level 2 (Follow-up) | Part 2b: VH4011499 Pre-specified Dose (Follow-up) | Matching Placebo for VH4011499 (Follow-up)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/3 | 0/7 | 0/6 | 0/7 | 0/3 | 0/6 | 0/6 | 0/6 | 0/3 | 0/7 | 0/6 | 0/7 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/3 | 0/7 | 0/6 | 0/7 | 0/3 | 0/6 | 0/6 | 0/6 | 0/3 | 0/7 | 0/6 | 0/7 | 0/3
Other Adverse Events (participants affected / at risk) | 3/6 | 2/6 | 2/6 | 2/3 | 2/7 | 4/6 | 2/7 | 1/3 | 1/6 | 3/6 | 4/6 | 1/3 | 3/7 | 3/6 | 5/7 | 0/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1a: VH4004280 Dose Level 1 (Monotherapy) (N=6) | Part 1a: VH4004280 Dose Level 2 (N=6) | Part 2a: VH4004280 Pre-specified Dose (Monotherapy) (N=6) | Matching Placebo for VH4004280 (Monotherapy) (N=3) | Part 1b: VH4011499 Dose Level 1 (Monotherapy) (N=7) | Part 1b: VH4011499 Dose Level 2 (Monotherapy) (N=6) | Part 2b: VH4011499 Pre-specified Dose (Monotherapy) (N=7) | Matching Placebo for VH4011499 (Monotherapy) (N=3) | Part 1a: VH4004280 Dose Level 1 (Follow-up) (N=6) | Part 1a: VH4004280 Dose Level 2 (Follow-up) (N=6) | Part 2a: VH4004280 Pre-specified Dose (Follow-up) (N=6) | Matching Placebo for VH4004280 (Follow-up) (N=3) | Part 1b: VH4011499 Dose Level 1 (Follow-up) (N=7) | Part 1b: VH4011499 Dose Level 2 (Follow-up) (N=6) | Part 2b: VH4011499 Pre-specified Dose (Follow-up) (N=7) | Matching Placebo for VH4011499 (Follow-up) (N=3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatophytosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
ViiV Healthcare agreements may vary with individual investigators, but will not prohibit any investigator from publishing. ViiV Healthcare supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT06039579/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT06039579/SAP_001.pdf